CLINICAL TRIAL: NCT05315349
Title: Retinal Microvascular Network and Coronary Revascularization Surgery at the Dijon University Hospital: Pilot Study
Brief Title: Retinal Microvascular Network and Coronary Revascularization Surgery at the Dijon University Hospital
Acronym: MRCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ARNOULD 2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Revascularization Surgery With Extracorporeal Circulation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient requiring cardiac surgery for myocardial revascularization (Experimental)
  Interventions: Other: Complete ophthalmological check-up; Biological: Blood sampling

INTERVENTIONS:
Other: Complete ophthalmological check-up — Preoperatively, 3 to 7 days after surgery and 1 to 2 months after surgery: fundus, optical coherence tomography angiography (OCT-A)
Biological: Blood sampling — Preoperatively and on Day 1 of surgery: 6 tubes of approximately 5 ml each, i.e. 30 ml

SUMMARY:
When coronary artery disease cannot be treated with medication, revascularization surgery can be performed. Although there have been many advances in recent years, this surgery is still associated with a high incidence of cardiovascular complications.

These complications are more frequent in patients with microscopic vessel damage. In clinical practice, microvascular status is difficult to characterize. Several models have been proposed, but they remain imprecise and are difficult to reproduce.

However, the study of the retinal microvascular network has recently emerged as a promising model. It is simple, quick and non-invasive thanks to the use of photographs or CT scans of the fundus (by optical coherence tomography angiography = OCT-A). Thus, the retinal vasculature is very often presented as an in vivo access that provides a window into systemic peripheral vasculature.

Despite the systematic assessment of cardiovascular risk by the usual risk factors (diabetes, hypertension, sex, etc.), risk stratification remains imperfect in coronary revascularization surgery and remains associated with a high incidence of complications, the most frequent being acute kidney injury (AKI).

Preoperative screening for retinal microvascular data could improve surgical risk stratification and better predict the potential occurrence of severe renal complications. Patient management could thus tailored to avoid such complications.

The main objective of the study is to investigate, in patients scheduled for coronary revascularization surgery with extracorporeal circulation, the discriminative capacity of retinal vascular density to predict the occurrence of AKI within 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who has given oral, free and informed consent
* Patient who is to undergo cardiac surgery for myocardial revascularization (coronary bypass surgery) with extracorporeal circulation at the Dijon University Hospital

Exclusion Criteria:

* Patient not covered by national health insurance
* Patient subject to a measure of legal protection (curatorship, guardianship)
* Acute circulatory collapse prior to surgery (amine, inotrope, circulatory assistance) preventing preoperative OCT-A
* Patient with macular disease (age-related macular degeneration, diabetic maculopathy, vascular occlusion)
* Pregnant, parturient or breastfeeding women
* Adult unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Failure (AKI) rate based on the Kidney Disease Improving Global Outcomes (KDIGO) Criteria | 7 days post-surgery
  Discriminative ability of mean retinal vascular density to predict acute kidney injury (defined by the KDIGO criteria) following coronary artery bypass grafting with extracorporeal circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No